CLINICAL TRIAL: NCT02925663
Title: Web-based Intervention to Improve Executive Functioning in Teens With Epilepsy (Epilepsy Journey)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21HD083335 (NIH)
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2018-07

CONDITIONS: Epilepsy
Keywords: executive functioning
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Patients are receiving an executive functioning intervention in an open trial design-pre-post
Oversight: Data Monitoring Committee: No

ARMS (1):
- EFI-E (Experimental): 10-session web-based modules to teach about executive functioning with videoconferencing with a therapist
  Interventions: Behavioral: EFI-E

INTERVENTIONS:
Behavioral: EFI-E — This is 10 web-based modules addressing foundational EF skills. Each online module will be accompanied by a videoconference with a therapist to review the skills and problem solve around adolescent-identified goals.

SUMMARY:
The purpose of this study is to establish the feasibility, accessibility, acceptability, and preliminary efficacy of an individually-tailored intervention to improve EF in adolescents with epilepsy (EFI-E).

DETAILED DESCRIPTION:
Epilepsy is a common childhood condition affecting approximately 326,000 youth in the United States. Adolescents with epilepsy are at significant risk for poor social and academic outcomes, neurobehavioral comorbidities (i.e., internalizing and externalizing symptoms), and poor treatment adherence. Studies have shown that one potential reason for these poor outcomes are deficits in executive functioning (EF), defined as the skills necessary for goal-directed and complex activities, including problem-solving, initiation, monitoring, organization, planning, self-regulation and working memory. EF deficits have been documented in 1/3 of youth with epilepsy, which is 3 times the prevalence in healthy youth. Evidence-based interventions to improve EF could play a critical role in preventing adverse outcomes (e.g., psychological comorbidities, non-adherence to the treatment regimen) and promoting optimal functioning in adolescents with epilepsy; however none exists for this vulnerable population. The aim of the current study is to establish the feasibility, accessibility, acceptability, and preliminary effects of an individually-tailored intervention to improve EF in adolescents with epilepsy (Executive Functioning Intervention-Epilepsy; EFI-E). Thirty participants will be recruited who have at least one clinically-elevated EF subscale or at least two at-risk subscale scores (> 1 standard deviation above the mean) on the parent Behavior Rating Inventory of Executive Function (BRIEF®)) to qualify for the EFI-E. EFI-E will consist of 10 web-based modules addressing foundational EF skills. Each online module will be accompanied by a videoconference with a therapist to review the skills and problem solve around adolescent-identified goals. Baseline and post-treatment questionnaires will be completed by adolescents and primary caregivers and electronically-monitored adherence will be obtained throughout the open trial. Participants will be in the trial for 9 months.

ELIGIBILITY:
Inclusion criteria

* Age 13-17 years
* Diagnosis of epilepsy
* Have at least two subclinical (>1 SD; T score between 60-65) or one clinically-elevated BRIEF subscale (T score > 65)
* Primary caregiver consent and adolescent assent to participate in study

Exclusion criteria

* Diagnosis of non-epilepsy medical disorders requiring daily medications with the exception of asthma and/or allergies
* Diagnosis of significant developmental disorders (e.g. Autism)
* Inability to read and speak English due to the questionnaires and intervention only been developed in English
* Family lives greater than 100 miles away from CCHMC
* If patient is planning to wean from their antiepileptic medication within the next 6 months

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Executive functioning: Behavior Rating Inventory of Executive Function (BRIEF) | 3-months

SECONDARY OUTCOMES:
Adherence: SimpleMed Pillboxes or MEMS TrackCaps | 3-months
Quality of life: PedsQL Epilepsy Module | 3-months
Seizures | 3-months
  A combination of chart review and parent-report will be used to create a composite seizure presence/absence variable.

OTHER OUTCOMES:
Child behavioral and emotional functioning: Behavior Assessment Schedule for Children-2 | 3-months
Treatment Feasibility | 3-months
  Treatment Feasibility and Acceptability Questionnaire
Executive functioning-BRIEF | 5-months
Executive functioning-BRIEF | 8-months
Adherence-SImple Med Pillbox or MEMS TrackCaps | 8-months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gutierrez-Colina AM, Clifford L, Wade SL, Modi AC. Uncovering Key Elements of an Executive Functioning Intervention in Adolescents: Epilepsy Journey. Clin Pract Pediatr Psychol. 2022 Jun;10(2):150-163. doi: 10.1037/cpp0000410. Epub 2021 Sep 2. PMID 35873364